CLINICAL TRIAL: NCT00052351
Title: A Pilot Study Of Sequential Vaccinations With Recombinant Vaccinia-CEA(6D)-TRICOM, And Recombinant Fowlpox-CEA(6D)-TRICOM (B7.1/ICIAM-1/LFA-3) With Sargramostim (GM-CSF), In Conjunction With Standard Adjuvant Chemotherapy In High Risk Breast Cancer Patients Status Post Surgery With 4+ Or More Lymph Nodes And CEA Expressing Tumors
Brief Title: Vaccine Therapy Plus Sargramostim and Chemotherapy in Treating Women With Stage II or Stage III Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000258196; NCI-03-C-0005; NCI-5191; NCT00047398 (obsolete NCT alias)
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2003-05

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — sargramostim; Cyclophosphamide; Doxorubicin; Paclitaxel; Radiotherapy

INTERVENTIONS:
Biological: recombinant fowlpox-CEA(6D)/TRICOM vaccine
Biological: recombinant vaccinia-CEA(6D)-TRICOM vaccine
Biological: sargramostim
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: paclitaxel
Radiation: radiation therapy

SUMMARY:
RATIONALE: Vaccines made from a gene-modified virus may make the body build an immune response to kill tumor cells. Colony-stimulating factors such as sargramostim may increase the number of immune cells found in bone marrow or peripheral blood. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining vaccine therapy with sargramostim and chemotherapy may kill more tumor cells.

PURPOSE: Randomized clinical trial to study the effectiveness of vaccine therapy plus sargramostim and combination chemotherapy in treating women who have undergone surgery for stage II or stage III breast cancer that has spread to the lymph nodes.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the immunological effects of 2 different schedules of vaccinia-CEA-TRICOM vaccine, fowlpox-CEA-TRICOM vaccine, and sargramostim (GM-CSF) administered with standard adjuvant chemotherapy in women with high-risk stage II or III breast cancer.
* Compare the safety of these regimens in these patients.
* Determine the feasibility of obtaining determinations of CD4 response in patients treated with these regimens.
* Compare disease-free survival of patients treated with these regimens.

OUTLINE: This is a randomized study. Patients are randomized to 1 of 2 treatment arms.

* Vaccinia-CEA-TRICOM: Beginning 2-3 weeks after surgery and before initiation of standard adjuvant chemotherapy, all patients receive vaccinia-CEA-TRICOM vaccine subcutaneously (SC) on day 1 and sargramostim (GM-CSF) SC on days 1-4 of week 1.
* Fowlpox-CEA-TRICOM: Patients are treated on 1 of the following schedules:

  * Arm I: During chemotherapy, patients receive fowlpox-CEA-TRICOM vaccine SC on day 1 and GM-CSF SC on days 1-4 of weeks 2, 5, 8, 11, 14, 17, 20, and 23. After chemotherapy, patients receive additional vaccinations on weeks 26, 38, and 50.
  * Arm II: Prior to chemotherapy, patients receive fowlpox-CEA-TRICOM vaccine SC on day 1 and GM-CSF SC on days 1-4 of week 2. After chemotherapy, patients receive additional vaccinations on weeks 26, 38, and 50.
* Chemotherapy: Patients receive doxorubicin IV over 5-7 minutes and cyclophosphamide IV over 30 minutes on day 1 of weeks 3, 6, 9, and 12. Patients then receive paclitaxel IV over 3 hours on day 1 of weeks 15, 18, 21, and 24. Treatment continues in the absence of disease progression (after at least 1 course of chemotherapy) or unacceptable toxicity.
* Radiotherapy: Patients undergo radiotherapy during weeks 26-32 in the absence of disease progression.

Patients with hormone-receptor positive tumors receive oral tamoxifen for 5 years beginning on approximately week 32.

Patients are followed every 6 months for 5 years.

PROJECTED ACCRUAL: A total of 28 (14 per treatment arm) patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the breast

  * Stage II or III
  * At least 4 positive lymph nodes
  * No inflammatory ductal carcinoma
* No positive lymph nodes by immunohistochemistry only
* Carcinoembryonic antigen (CEA) expression, as indicated by 1 of the following:

  * At least 30% of tumor stains for CEA on immunohistochemistry
  * Elevated serum CEA (greater than 5 ng/mL) anytime during disease course
* Must be HLA-A2 positive
* Must have received prior vaccinia for smallpox immunization with 1 of the following as evidence:

  * If age 25 and under, physician certification of prior vaccination
  * If over age 25, patient recollection and vaccination-site scar
  * Any age, detectable anti-vaccinia antibodies
* No metastases by CT scan of chest, abdomen, and pelvis and a bone scan
* Hormone receptor status:

  * Estrogen receptor status and progesterone receptor status known

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Menopausal status:

* Not specified

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT and SGPT no greater than 1.5 times ULN
* Hepatitis B and C negative

Renal

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance greater than 60 mL/min
* No proteinuria OR
* Protein less than 1,000 mg per 24-hour urine collection
* No hematuria
* No abnormal sediment

Cardiovascular

* LVEF at least 45% by echocardiogram or MUGA if either of the following are true:

  * History of cardiac disease
  * Received prior cardiotoxic chemotherapy

Immunologic

* No evidence of immunocompromised status
* No autoimmune disease such as any of the following:

  * Autoimmune neutropenia, thrombocytopenia, or hemolytic anemia
  * Systemic lupus erythematosus
  * Sjogren's syndrome
  * Scleroderma
  * Myasthenia gravis
  * Goodpasture syndrome
  * Addison's disease
  * Hashimoto's thyroiditis
  * Active Graves' disease
* No active or prior eczema or other eczematoid skin disorders
* No other acute, chronic, or exfoliative skin conditions (e.g., atopic dermatitis, burns, impetigo, varicella zoster, severe acne, or other open rashes or wounds)
* HIV negative
* No active infection within the past 3 days
* No allergy to eggs
* No history of allergy or untoward reaction to prior vaccination with vaccinia virus

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other serious illness
* No other malignancy within the past 3 years except squamous cell or basal cell skin cancer
* No history of seizures, encephalitis, or multiple sclerosis
* No active inflammatory bowel disease
* Must be able to avoid close household contact with the following during and for 2 weeks after vaccinations:

  * Persons with active or prior eczema or other eczematoid skin disorders
  * Persons with any other acute, chronic, or exfoliative skin conditions (e.g., atopic dermatitis, burns, impetigo, varicella zoster, severe acne, or other open rashes or wounds)
  * Pregnant or nursing women
  * Children under 5 years old
  * Immunodeficient or immunosuppressed persons (by disease or therapy), including those with HIV infection

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics

Chemotherapy

* No prior doxorubicin, cyclophosphamide, or paclitaxel

Endocrine therapy

* No concurrent steroids except the following:

  * Topical steroids
  * Inhaled steroids for moderate asthma
  * Dexamethasone prior to taxanes

Radiotherapy

* No prior radiotherapy to more than 50% of the lymph nodes

Surgery

* At least 2 weeks since prior surgery and recovered
* No prior splenectomy

Other

* No other concurrent anti-tumor therapies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-09; Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip M. Arlen, MD, Study Chair — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - Center for Cancer Research, Bethesda, Maryland